CLINICAL TRIAL: NCT06907394
Title: Effect of Osteopathic Manipulations of Post Cesarean Section Adhesions on Low Back Pain
Brief Title: Osteopathy of Post Cesarean Section Adhesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adly A Adam (Other)
Responsible Party: Sponsor-Investigator, Adly A Adam, Lecturer of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003148
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Cesarean Section Complications
Keywords: Osteopathic Manipulation; Low Back Pain; Post Cesarean Section Adhesions; Visual Analogue Scale; Oswestry Low Back Disability Questionnaire; Modified Schober Test
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, Pre/Posttreatment, Controlled Trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The whole participants, care provider, investigator and the outcome assessor will not be aware of each participant allocation within the current study groups; Based on a third person will be assigned for randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Fifteen Females will receive only analgesic drugs for four weeks.
  Interventions: Other: Control Group
- Study Group (Experimental): Fifteen females will receive osteopathic manipulations once weekly along four weeks, plus analgesic drugs for four weeks.
  Interventions: Other: Osteopathic Manipulations; Other: Control Group

INTERVENTIONS:
Other: Osteopathic Manipulations — Osteopathic Manipulations (a. Myofascial release technique: Direct scar release+ Indirect scar release 'Fascial unwinding'; b. Grand Maneuver; Visceral manipulations of uterus
  Arms: Study Group
Other: Control Group — Paracetamol tablets

SUMMARY:
Chronic low back pain post cesarean section adhesions represents a restricting dysfunction, mainly influences abdominal fascia that leads to major welfare and economic restrictions. Osteopathic manipulation is a drug-free non-invasive is the therapeutic application of manually guided forces to improve physiologic function and support homeostasis. The purpose of the current study is to determine the effect of osteopathic manipulations of post cesarean section adhesions on low back pain

DETAILED DESCRIPTION:
Chronic low back pain is a common musculoskeletal disorder affects adults with 84% prevalence. It influences lower back, and lasts at least 12 weeks. Where increased annual cesarean section rates up to 19.1% associated with scar, pelvic, abdominal and low back pain disorders (Chia et al., 2016). From the fascial point of view, abdominal muscles are in continuity with the thoracolumbar fascia and the pelvic floor. It has been demonstrated that they work with great synergy and guaranteed by fascial continuity (Fan et al., 2018).

Osteopathic manipulative technique consists of a range of direct, indirect, combined, fluid and reflex-based manual techniques that are applied specifically to a joint or non-specifically to a body area. Direct techniques apply thrust, impulse, muscle contraction, fascial loading or passive range of motion (Fan et al., 2018).The purpose of the current study is to determine the effect of osteopathic manipulations of post cesarean section adhesions on low back pain. Up on that 30 post cesarean women suffering from low back pain at least for 6 months from the Outpatient Clinic of Mitghamer Hospital, El-Daqahlia. Their age range 20-35 years old, BMI range≤ 25 kg /m2. They will be allocated into control group will receive analgesics. Study group will receive four weeks of analgesics, plus osteopathic manipulations once per week.

ELIGIBILITY:
Inclusion Criteria:

* They suffered from low back pain and undergoes cesarean section at least 6 months before entry into study.
* Their body mass index (BMI) will be ≤ 25 kg /m2.
* Their age will range from 20 to 35 years.
* They would not use any other analgesic drugs during the study period.

Exclusion Criteria:

* Pregnancy or suspected pregnancy.
* Recent abdominal surgery
* Patients with severe spinal pathology (cauda equine syndrome, spinal canal stenosis, fracture of spine, discitis, infectious disease of spine).
* Cancer.
* Abdominal and pelvic infection, open wound, burn and skin irritation.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study targeting post cesarean section adhesions (among women) on low back pain management.
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Baseline, and Post-treatment of the the study treatment program along 4-weeks).
  a self-reported pain measurement a widely utilized scale in rehabilitation. It has been shown to be valid and reliable, and its ratio scale properties make VAS the optional tool for describing pain intensity

SECONDARY OUTCOMES:
Oswestry Low Back Disability Questionnaire | Baseline, and Post-treatment of the the study treatment program along 4-weeks).
  An extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. It consists of 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability). Each question is scored from 0-5 (minimum to maximum).The point total from each section is summed and the then divided by the total number of questions answered and multiplied by 100 to create a percentage disability. The scores range from 0-100% with lower scores meaning less disability.
Modified Schober Test | Baseline, and Post-treatment of the the study treatment program along 4-weeks).
  The Modified Schober test is designed to measure the range of lumbar flexion in patients. The positive Schober test result is when the distance between the two lines does not increase by at least 5cm when the person bends forward. The normative values were found to be 6.85 ±1.18 cm for flexion, and 2.42±0.74 cm for extension.

CONTACTS AND LOCATIONS:
Overall Officials: Khadija S Abdulaziz, PHD, Study Chair — Professor of Physical Therapy for Woman's Health; Mohamed A Abo Elainin, PHD, Study Director — Consultant of Obstetrics and Gynecology
Locations (1):
- Mitghamer Hospital, Mitghamer city, Qalyubia Governate, Al Maţmar, Qalubyia, Egypt

IPD SHARING:
Plan to Share IPD: No